CLINICAL TRIAL: NCT04282356
Title: Intensive Intraperitoneal Therapy in Advanced Ovarian Cancer Combining Cytoreductive Surgery With Hyperthermic Intraperitoneal Chemotherapy (HIPEC) and Postoperative Intraperitoneal Chemotherapy (IPC)
Brief Title: Intensive Intraperitoneal Therapy in Advanced Ovarian Cancer
Acronym: INTENS-IP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROICM 2019-08 INT
Record Dates: First submitted 2020-01-08; First posted 2020-02-24 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Cancer; Intraperitoneal Chemotherapy
Keywords: ovarian cancer; intraperitoneal; chemotherapy; surgery; HIPEC
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraperitoneal chemotherapy (Experimental): Cisplatin 100mg/m2 during surgery IV Paclitaxel, 135mg/m2 on D1, IP Carboplatin, AUC 6 on D1, and IP Paclitaxel, 60mg/m2 on D8 after surgery with at least 3 courses performed (up to 4-6 allowed)
  Interventions: Drug: Intraperitoneal chemotherapy during surgery

INTERVENTIONS:
Drug: Intraperitoneal chemotherapy during surgery — During interval surgery the patient will undergo HIPEC (Cisplatin 100mg/m2, 1h 30 infusions with sodium thiosulfate renal protection). They will then receive postoperative IPC i.e intravenous and intraperitoneal administration (IV Paclitaxel, 135mg/m2 on D1, IP Carboplatin, AUC 6 on D1, and IP Paclitaxel, 60mg/m2 on D8) with at least 3 courses performed (up to 4-6 allowed).
  Other Names: Intraperitoneal chemotherapy after surgery

SUMMARY:
Clinicians postulate that it may be interesting to combine the two IntraPeritoneal (IP) treatments associated with a significant improvement of OC overall survival i.e. cytoreductive surgery with hyperthermic intraperitoneal chemotherapy (HIPEC) and postoperative intraperitoneal chemotherapy (IPC) as an " intensive peritoneal " regimen in the initial management of stages III-IVA ovarian cancers. Performing a postoperative IPC may allow completing and extending the duration of the effect of HIPEC in decreasing the risk of peritoneal recurrence. HIPEC may also allow administering an early IP treatment on the residual microscopic disease during initial or interval surgery with an optimal access to the intraperitoneal cavity. Postoperative IPC will extend the HIPEC effect on unsterilized peritoneal microscopic residues with the aim of decreasing the risk of local recurrence. Performing HIPEC before IPC could allow limiting the number of postoperative IP courses needed. Nevertheless, this association questions its feasibility and tolerance, which should both be assessed in a phase II trial. Clinicians propose to conduct this feasibility study combining for the first time HIPEC with IPC as first-line treatment of ovarian cancer with peritoneal carcinomatosis to perform a peritoneal intensification.

DETAILED DESCRIPTION:
Epithelial ovarian cancer (EOC) is the main cause of gynecological cancer death in developed countries, reflecting a clinical diagnosis possible at an advanced-stage of the disease and an early propensity for peritoneal dissemination. The treatment of these advanced stages combines optimal cytoreductive surgery and a platinum and taxan-based systemic chemotherapy. Despite a very high initial chemosensitivity and frequent clinical complete responses, the majority of patients relapses after a mean period of 18 months and progressively develops resistance to the various chemotherapeutic treatments. Nevertheless, recurrences remain frequently located in the peritoneal cavity.

Intraperitoneal administration of chemotherapeutic agents (intraperitoneal chemotherapy, IPC) is adapted to OC natural history. IPC has shown its clinical efficacy compared with intravenous (IV) chemotherapy in three randomized clinical trials. Recently, an unexpected median overall survival of 110 months was reported after complete surgery followed with IPC. Nevertheless, IPC repetitions are still strongly limited due to the high local toxicities and the difficult access to the peritoneal cavity leading to an important morbidity of the IP catheters. In the GOG-172 trial, half of the patients of the IPC arm did not receive the complete planned IP treatment. Long-term results of both the GOG-172 and GOG-114 trials showed that treatment efficacy is correlated with the numbers of IPC courses administered and with a significant long-term effect for patients receiving 3 or more IPC courses. For patients receiving neoadjuvant chemotherapy and optimal debulking surgery, the OV21 study recently showed that IP carboplatin-based chemotherapy was well tolerated and associated with an improved disease-free survival rate at 9 months after surgery compared with that of the IV chemotherapy group.

At the same time, complete cytoreductive surgery associated with perioperative hyperthermic intraperitoneal chemotherapy (i.e. HIPEC) is the second promising IP treatment that is currently evaluated in advanced OC. HIPEC allows an early IP treatment enhanced by hyperthermia while limiting the diffusion problem of the IP drugs and the difficult access to the peritoneal cavity. Nevertheless, despite this promising concept, HIPEC with a unique and limited IP cisplatin dose remains discussed in the management of OC. A phase 3 trial (OVHIPEC study), recently published in the New England Journal of Medicine, emphasized the therapeutic interest of a cisplatin-based HIPEC procedure at the time of interval surgery for patients receiving neoadjuvant chemotherapy. A significant improvement of overall survival (12 months gain: OS 33.9 months vs 45.7 months for IDS with HIPEC HR = 0.67 (0,48-0,94) p=0,02) was demonstrated for patients receiving HIPEC with a favorable tolerance profile and no additional morbidity.

Clinicians postulate that it may be interesting to combine the two IP treatments associated with a significant improvement of OC overall survival i.e. cytoreductive surgery with HIPEC and postoperative IPC as an " intensive peritoneal " regimen in the initial management of stages III-IVA ovarian cancers. Performing a postoperative IPC may allow completing and extending the duration of the effect of HIPEC in decreasing the risk of peritoneal recurrence. HIPEC may also allow administering an early IP treatment on the residual microscopic disease during initial or interval surgery with an optimal access to the intraperitoneal cavity. Postoperative IPC will extend the HIPEC effect on unsterilized peritoneal microscopic residues with the aim of decreasing the risk of local recurrence. Performing HIPEC before IPC could allow limiting the number of postoperative IP courses needed. Nevertheless, this association questions its feasibility and tolerance, which should both be assessed in a phase II trial. Clinicians propose to conduct this feasibility study combining for the first time HIPEC with IPC as first-line treatment of ovarian cancer with peritoneal carcinomatosis to perform a peritoneal intensification.

Design:

After written informed consent, patients presenting with suspected advanced OC will undergo an exploratory laparoscopy with biopsies and evaluation of the disease extent (Sugarbaker PCI score). Only patients with histologically-proven high-grade serous OC with extended disease (stages III B-C and IV-A with minimal pleural effusion (FIGO 2014) will be included in the study. Patients with stage IV-A cancer with major pleural effusion and stage IV-B patients will be excluded. Patients with extended peritoneal carcinomatosis considered unresectable at exploratory laparoscopy will undergo classical 3-4 courses neoadjuvant chemotherapy followed by interval surgery and will be selected to participate to the INTENSIP study.

During interval surgery, patients who will have undergone complete surgery (no macroscopic residue) and who gave their written consent will be included and will undergo HIPEC (Cisplatin 100mg/m2, 1h 30 infusions with sodium thiosulfate renal protection).

They will then receive postoperative IPC i.e intravenous and intraperitoneal administration (IV Paclitaxel, 135mg/m2 on D1, IP Carboplatin, AUC 6 on D1, and IP Paclitaxel, 60mg/m2 on D8) with at least 3 courses performed (up to 4-6 allowed, depending on the classical therapeutic strategy of each participating center). In case of toxicity or inability to administer the treatment in an IP manner, it will be given intravenously.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75 years,
* Patients with high-grade serous (high grade according to MD Anderson, grade II and III according to Silverman) ovarian or tubal or primitive peritoneal histologically proven cancer,
* Initial laparoscopy confirming the histological type, evaluating the extent of the disease by PCI score and confirming the initial non-resectability,
* Stage III B-C (FIGO 2014) or stage IVA with minimal or moderate pleural effusion (measured on a thoracic CT scanner, the largest thickness of which is less than 3 cm),
* Complete interval cytoreduction surgery,
* Indication of 3 to 4 cures of neoadjuvant chemotherapy based on the Carboplatin-Paclitaxel (carbo-taxol) combination,
* The delay between the last course of NAT and the surgery must be between 4 and 8 weeks,
* Hematologic function, hemoglobin ≥ 10 g / dl; PNN ≥ 1 x 109 / L, platelets ≥ 100 x 109 / L,
* Total bilirubin ≤ 1.5 LSN, ALT or AST ≤ 3 ULN,
* Absence of renal insufficiency (creatinine clearance ≤ 70 ml / min) according to the MDRD method,
* Informed consent signed before any specific procedure under consideration,
* Patients affiliated to the French social security scheme or equivalent.

Exclusion Criteria:

* Performance Index (WHO) ≥ 2,
* Stage IV B or IV A with significant pleural effusion (measured on a thoracic CT scanner, the largest thickness of which is more than 3 cm),
* Renal impairment (clearance <70 ml / min) according to the MDRD method,
* General contraindication to the realization of a tumor reduction surgery or HIPEC (contraindication or history allergic reaction to any treatments components),
* Hepatic insufficiency (bilirubin > 1.5 x normal, ASAT & ALAT > 3 x upper limit of normal),
* Serious life-threatening co-existing condition at stake,
* Cardio-respiratory pathology indicating hyper hydration, to be implemented for HIPEC,
* Patient who has already been treated with chemo-hyperthermia for ovarian cancer,
* History of cancer, except basal cell carcinoma of the skin or carcinoma in situ of cervix having recurred within five years prior to entry into this trial,
* Any severe untreated infectious disease,
* Peripheral sensory neuropathy ≥ grade 2 at the inclusion time,
* Patients whose regular follow-up is a priori impossible for psychological, family, social or geographical reasons,
* Pregnant and / or nursing women,
* Subjects under tutelage, curatorship or safeguard of justice.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
The success of the combination of HIPEC and IPC assessed by chemotherapy administration after surgery | Until the chemotherapy courses completion: 6 months after interval surgery
  Number of administred courses of intraperitoneal chemotherapy during the 6 months following complete interval cytoreductive surgery with HIPEC.
The success of HIPEC and IPC combination assessed by surveillance safety | Until the chemotherapy courses completion: 6 months after interval surgery
  Rate of HIPEC tolerance (deterioration of the renal function and morbidity of HIVEC) and CIP tolerance (abdomibal pain and complications of the IP treatment)

SECONDARY OUTCOMES:
Morbidity rate of reductive surgery combined with HIPEC according to the CLAVIEN and DINDO score | Up to 60 postoperative days
  Morbidity rate according to the CLAVIEN and DINDO score
HIPEC toxicities | 2 months after interval surgery
  according to the CTC-AE v5.0 scale
IPC toxicities | Until the chemotherapy courses completion: 6 months after interval surgery
  according to the CTC-AE v5.0 scale
Complications | after interval surgery with HIPE: 2 months
  Complications due to intraperitoneal catheters
Relapse-Free survival | Until study completion: 5 years
  Relapse Free Survival is defined as the time from the date of inclusion to first documentation of objective tumor progression or to death due to progression

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ROUANET, MD, Study Chair — Institut Régional du Cancer de Montpellier (ICM)
Locations (1):
- Institut du Cancer de Montpellier - Val d'Aurelle, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cannistra SA. Cancer of the ovary. N Engl J Med. 2004 Dec 9;351(24):2519-29. doi: 10.1056/NEJMra041842. No abstract available. PMID 15590954
- [Background] Colombo PE, Mourregot A, Fabbro M, Gutowski M, Saint-Aubert B, Quenet F, Gourgou S, Rouanet P. Aggressive surgical strategies in advanced ovarian cancer: a monocentric study of 203 stage IIIC and IV patients. Eur J Surg Oncol. 2009 Feb;35(2):135-43. doi: 10.1016/j.ejso.2008.01.005. Epub 2008 Mar 4. PMID 18289825
- [Background] Armstrong DK, Bundy B, Wenzel L, Huang HQ, Baergen R, Lele S, Copeland LJ, Walker JL, Burger RA; Gynecologic Oncology Group. Intraperitoneal cisplatin and paclitaxel in ovarian cancer. N Engl J Med. 2006 Jan 5;354(1):34-43. doi: 10.1056/NEJMoa052985. PMID 16394300
- [Background] van Driel WJ, Koole SN, Sikorska K, Schagen van Leeuwen JH, Schreuder HWR, Hermans RHM, de Hingh IHJT, van der Velden J, Arts HJ, Massuger LFAG, Aalbers AGJ, Verwaal VJ, Kieffer JM, Van de Vijver KK, van Tinteren H, Aaronson NK, Sonke GS. Hyperthermic Intraperitoneal Chemotherapy in Ovarian Cancer. N Engl J Med. 2018 Jan 18;378(3):230-240. doi: 10.1056/NEJMoa1708618. PMID 29342393